CLINICAL TRIAL: NCT02852265
Title: Nexplanon Use in Women Primarily Choosing a Combined Hormonal Contraceptive: a Proof of Concept Trial
Brief Title: Nexplanon and Combined Oral Contraceptive (COC) Combined Use Study
Acronym: NexTOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 890433
Record Dates: First submitted 2016-07-13; First posted 2016-08-02 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Contraception
Keywords: oral contraceptive; contraceptive implant; contraception; adherence; adverse event
MeSH Terms: interventions — etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COC users or new starts (Experimental): Subjects will have a etonogestrel contraceptive implant placed at enrollment. Women using COC as method of contraception for at least 1 month will be considered COC users. Women starting a COC or recently started a COC within the past month will be considered new starts.
  Interventions: Drug: Etonogestrel contraceptive implant

INTERVENTIONS:
Drug: Etonogestrel contraceptive implant — Place nexplanon
  Other Names: Nexplanon

SUMMARY:
Women currently using or starting a combined oral contraceptive will be offered study enrollment. Study subjects will have a Nexplanon placed and followed for 6 months to evaluate if they continue the COC, continue the implant, or both, and to assess adverse events and bleeding patterns.

DETAILED DESCRIPTION:
The investigators will recruit women being seen in a UC Davis medical office or who contact our research office. Potential participants must be women currently COCs or intending to initiate COCs at the time of the office visit. The investigators expect that most women will be recruited while in the office who decide to initiate COCs or are continuing COC use-these women will be offered the ability to talk to research staff about the study.

Visit 1:

Informed consent will be obtained. As part of informed consent, subjects will be educated that there is little data available on the adverse effects of combined COC and ENG implant use. The consent form will include a standardized description of the side effects and bleeding profile of COCs and the implant. Subjects will also need to review the package label information for Nexplanon and sign the FDA-required Nexplanon consent. After obtaining informed consent, subjects will be screened for entry criteria. Medical history will be obtained. A urine pregnancy test will be performed. Eligible subjects will receive a prescription for the desired COC (if needed) and have a Nexplanon contraceptive implant placed. A diary will be dispensed for the subject to document daily bleeding, COC use and adverse events.

Follow-up A follow-up visit will occur at 1 month (+1 week) and 3 and 6 months (+2 weeks). The diary will be reviewed and a copy made to keep with the source documentation. Adverse events will be determined by inquiry and diary review. The subject will inform the study staff if she is using her COC and if she wants to continue use of her COC and ENG implant. At the 1 and 3 month visits, additional diaries will be dispensed as needed. The ENG implant will be removed upon request at any time during the study.

A phone call will occur approximately 1 week prior to the 3 and 6 month visits to check status and remind subject of the scheduled visit. Study participation will be complete after the 6 month follow-up visit.

No surveys will be used that the subject fills out herself. A daily diary will be used.

No blood draws will occur during this study.

Data to be collected by study staff include demographics, past medical and gynecologic history, prior and current contraceptive use, and reason for using COC (contraception, medical or both).

Because women are being enrolled who are already currently using COCs or who plan to start COCs, the COC is not a study drug. The study intervention (study drug) is the contraceptive implant. The systemic hormone exposure with a contraceptive implant is minimal relative to a COC. We would not expect any increase in side effects by adding a contraceptive implant to COC users. Of note, the primary risk with COC use is related to the estrogen which can increase the risk of venous thromboembolic disease. The implant has no estrogen. All products being used in the study are FDA-approved for contraception.

ELIGIBILITY:
Inclusion:

* Women being seen in a UC Davis medical office or who contact our research office.
* Potential participants must be women currently COCs or intending to initiate COCs at the time of the office visit.

Exclusion:

* Women who have contraindications to using a COC or a contraceptive implant (Category 3 or 4 in the CDC Medical Eligibility Criteria) will be excluded.
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Creinin, MD, Principal Investigator — Univeristy of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MJ, Hsia JK, Creinin MD. Etonogestrel implant use in women primarily choosing a combined oral contraceptive pill: A proof-of-concept trial. Contraception. 2018 Jun;97(6):533-537. doi: 10.1016/j.contraception.2018.02.009. Epub 2018 Feb 26. PMID 29496473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We consented and enrolled 20 women in the outpatient clinic at the University of California, Davis Department of Obstetrics and Gynecology for study participation between September and December 2016.
Groups:
- New Start COC Users: Women who are starting or recently started (within last 4 weeks) a combined oral contraceptive
- Continuing COC Users: Women who have been using a combined oral contraceptive for more than 4 weeks
Period: 1-month Follow-up
Arm/Group | New Start COC Users | Continuing COC Users
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: 3-month Follow-up
Arm/Group | New Start COC Users | Continuing COC Users
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: 6-month Follow-up
Arm/Group | New Start COC Users | Continuing COC Users
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- New Start COC Starters: Women who are starting or recently started (within last 4 weeks) a combined oral contraceptive
- Total: Total of all reporting groups
Arm/Group | New Start COC Starters | Continuing COC Users | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 25 [20 to 34] | 20.5 [16 to 34] | 23 [16 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 6 | 5 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Pill type [Count of Participants; unit: Participants]
  21/7 monophasic | 7 | 5 | 12
  24/4 monophasic | 0 | 1 | 1
  21/7 triphasic | 1 | 2 | 3
  Continuous dosing | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluating ENG as Acceptable: Acceptability (Measurement: Questionnaire)
Description: Evaluate the acceptability (continuation of the implant throughout the study) of concomitant etonogestrel (ENG) implant use in women choosing a combined oral contraceptive (COC) for contraception
Time Frame: 6 months
Population: All women enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | New Start COC Users | Continuing COC Users
Number analyzed (Participants) | 10 | 10
Participants | 9 | 8

2. Primary Outcome: Number of Participants Evaluating ENG as Tolerable: Tolerability (Measurement: Diaries and Questionnaire)
Description: Evaluate the tolerability (side effects) of concomitant etonogestrel (ENG) implant use in women choosing a combined oral contraceptive (COC) for contraception
Time Frame: 6 months
Population: All enrolled subjects, new or worsening side effects after 6 months of use in women using both an implant and a COC
Measure: Number; unit: participants
Arm/Group | New Start COC Users | Continuing COC Users
Number analyzed (Participants) | 5 | 5
participants
  headache | 2 | 0
  nausea | 1 | 0
  mastalgia | 1 | 0
  mood complaints | 1 | 0
  worsening acne | 2 | 0
  worsening dysmenorrhea | 2 | 1
  weight gain | 2 | 1

3. Secondary Outcome: Patient Interest (Measurement: Ability to Enroll)
Description: Demonstrate that women desiring a COC are willing to use ENG implant concomitantly as a continuous "back-up" contraceptive
Time Frame: 6 months
Population: women using or starting a COC and having an etonogestrel implant placed; 1 lost to follow-up in each group from enrollment (n=10 in both groups at enrollment)
Measure: Count of Participants; unit: Participants
Groups:
- COC Users: Subjects will have a etonogestrel contraceptive implant placed at enrollment. Women using COC as method of contraception for at least 1 month will be considered COC users.
- COC New Starts: Subjects will have a etonogestrel contraceptive implant placed at enrollment. Women starting a COC or recently started a COC within the past month will be considered new starts.
Arm/Group | COC Users | COC New Starts
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

4. Secondary Outcome: Bleeding Patterns (Measurement: Diaries)
Description: Bleeding patterns while using a COC concomitantly with ENG implant
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- COC Users: Subjects will have a etonogestrel contraceptive implant placed at enrollment. Women using COC as method of contraception for at least 1 month will be considered COC users.
  Etonogestrel contraceptive implant: Place nexplanon
- New Starts: Subjects will have a etonogestrel contraceptive implant placed at enrollment. Women starting a COC or recently started a COC within the past month will be considered new starts.
  Etonogestrel contraceptive implant: Place nexplanon
Arm/Group | COC Users | New Starts
Number analyzed (Participants) | 9 | 9
Participants
  prolonged 1st 90 days | 1 | 1
  frequent 1st 90 days | 2 | 1
  irregular 1st 90 days | 2 | 2
  infrequent 1st 90 days | 1 | 3
  amenorrhea 1st 90 days | 0 | 0
  regular 1st 90 days | 3 | 2
  prolonged 2nd 90 days | 0 | 1
  frequent 2nd 90 days | 0 | 2
  irregular 2nd 90 days | 2 | 2
  infrequent 2nd 90 days | 5 | 2
  amenorrhea 2nd 90 days | 1 | 1
  regular 2nd 90 days | 1 | 1

5. Secondary Outcome: COC Continuation Rate (Measurement: Participant Interview)
Description: Continuation rate of COC over 6 months of evaluation regardless on whether or not the implant was still present at 6 months
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COC Users | New Starts
Number analyzed (Participants) | 9 | 9
Participants | 6 | 5

6. Secondary Outcome: Post-study Method Plan (Measurement: Participant Interview)
Description: Plan to continue the COC and/or implant after the study based on interview at last visit
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COC Users | New Starts
Number analyzed (Participants) | 9 | 9
Participants
  using implant only | 3 | 4
  using COC only | 1 | 3
  using implant and COC | 5 | 2
  not using implant or COC | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months of follow-up
Arm/Group | New Start COC Users | Continuing COC Users
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Start COC Users (N=10) | Continuing COC Users (N=10)
Nexplanon removal (Surgical and medical procedures) | 1 (1) | 1 (1) — removal of implant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT02852265/Prot_SAP_000.pdf